CLINICAL TRIAL: NCT01740895
Title: A Prospective, Observational, Non-randomized, Double Blind, Global, Multi-center Registry With an Adaptive Design, Investigating the Diagnostic Utility of Instantaneous Wave-free Ratio™ (iFR®) in Assessing Coronary Stenosis Relevance.
Brief Title: ADenosine Vasodilator Independent Stenosis Evaluation II - ADVISE II
Acronym: ADVISEII
Status: Completed | Type: Observational
Sponsor: Volcano Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: PFC-001
Record Dates: First submitted 2012-11-16; First posted 2012-12-04 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To assess the clinical value of iFR to characterize, without concomitant administration of hyperemic agents and outside a specified range of iFR values, coronary stenosis severity as determined with fractional flow reserve (FFR)

ELIGIBILITY:
Inclusion Criteria:

* - Patient must be > 18 and < 85 years of age
* Willing to participate and able to understand, read and sign the informed consent document before the planned procedure
* Eligible for coronary angiography and/or percutaneous coronary intervention
* Coronary artery disease with at least 1 or more visually assessed coronary stenoses (>40% diameter stenosis) in native major epicardial vessel or its branches by coronary angiogram.
* Stable angina or acute coronary syndromes (non-culprit vessels only and outside of primary intervention during acute myocardial infarction)

Exclusion Criteria:

* - Known contraindication to adenosine administration
* Implanted temporary or permanent artificial pacemakers, Left Bundle Branch Block (LBBB), 1st and 2nd degree AV Block
* STEMI or non STEMI within 48 hours of procedure
* Any contraindications for FFR interrogation or percutaneous coronary intervention (PCI) as determined by the investigator
* Severe vessel tortuosity and/or severe calcification by angiogram
* Significant valvular pathology (moderate or severe AS/AR/MS/MR)
* Previous Coronary Artery Bypass surgery with patent grafts to the interrogated vessel
* Weight >200kg (441 lbs.)
* Hemodynamic instability at the time of intervention (heart rate<50 beats per minute, systolic blood pressure <90mmHg) balloon pump
* Significant hepatic disease, renal disease, lung disease (pulmonary chronic pulmonary obstructive disease) and/or malignant disease with unfavorable prognosis or presenting with abnormal serum laboratory values that the physician believes is clinically significant
* Contraindication to antithrombotic regimen or anticoagulation therapy
* History of or known reaction or sensitivity to contrast agent and is unable to be pre-medicated
* Left main stenosis, tandem stenosis separated by more than 5 mm that require separate pressure guide wire interrogation or PCI (not to be interrogated or treated as a single stenosis), or total occlusions
* Known Left ventricular ejection fraction (LVEF) <30%

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient receiving a standard of care FFR measurment in the cath lab setting.
Sampling Method: Non-Probability Sample
Enrollment: 818 (Actual)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Hemodynamic Severity | at the time of study procedure- 1 day
  Percentage of stenosis properly classified in terms of hemodynamic severity by iFR values ≤0.85 and ≥0.94. Hemodynamic severity will be established with an FFR value ≤ 0.80.

SECONDARY OUTCOMES:
Specificity | at the time of study procedure- 1 day
  Minimum iFR exclusion ranges around iFR 0.89 in which iFR and FFR agreement is equal to or greater than 80% and 90%

OTHER OUTCOMES:
Sensitivity | at the time of study procedure- 1 day
  Minimum iFR exclusion ranges around iFR 0.89 in which iFR and FFR agreement is equal to or greater than 80% and 90%

CONTACTS AND LOCATIONS:
Overall Officials: Javier Escaned, MD, Principal Investigator — Hospital Cl¡nico San Carlos Madrid Spain; Amir Lerman, MD, Principal Investigator — Mayo Clinic Rochester MN USA
Locations (44):
- United States (30):
  - Chandler Regional Medical Center, Chandler, Arizona
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - Coloado Heart and Vascular/St Anthony's, Lakewood, Colorado
  - Cardiovascular Research of Florida, Gainesville, Florida
  - North Florida regional Medical center, Gainsville, Florida
  - Baptist Cardiac & Vascular Institute, Miami, Florida
  - Winter Haven Hospital, Winter Haven, Florida
  - St Johns Hospital/ Prairie Education and Research, Springfield, Illinois
  - University of Minnesota, Minneapolis, Minnesota
  - St. Marys Hospital/ MAYO Clinic, Rochester, Minnesota
  - Regions Hospital Heart Center, Saint Paul, Minnesota
  - Washington University, St Louis, Missouri
  - AtlantiCare Regional Medical Center, Pomona, New Jersey
  - Stony Brook Medicine, Stony Brook, New York
  - University of North Carolina Hospital, Chapel Hill, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - East Carolina University/ Pitt County Hospital, Greenville, North Carolina
  - Wake Heart research/ Rex Hospital, Raleigh, North Carolina
  - Wake Heart research/ Wake Medical Center, Raleigh, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Geisinger Medical Center, Danville, Pennsylvania
  - UPMC Hamot, Erie, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Allegheny General, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - VA Charleston (RALPH H. JOHNSON VA MEDICAL CENTER), Charleston, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Wellmont Holston Valley Medical center, Kingsport, Tennessee
  - Sentara Health/Norfolk General Hospital, Norfolk, Virginia
  - Auora St Lukes, Milwaukee, Wisconsin
- Victoria Heart Institute Foundation, Victoria, British Columbia, Canada
- Al Dorrah, Cairo, Egypt
- Kerckhoff Klinik Bad Nauheim, Bad Nauheim, Germany
- Netherlands (4):
  - AMC Amsterdam, Amsterdam
  - Breda Amphia Ziekenhuis, Breda
  - Medische Spectrum Twente, Enschede
  - ERASMUS MC Rotterdam, Rotterdam
- Poland (3):
  - Jagiellonian University, Institute of Cardiology, Krakow
  - MSWiA Warszawa Woloska, Warsaw
  - Polikliniką SP ZOZ we Wrocławiu, Wroclaw
- Spain (3):
  - Hospital Universitario San Juan, Alicante
  - Hospital Universitario La Paz de Madrid, Madrid
  - Hospital Cl¡nico San Carlos, Marid
- Liverpool Heart and Chest Hospital, Liverpool, United Kingdom

REFERENCES:
- [Derived] Echavarria-Pinto M, van de Hoef TP, Garcia-Garcia HM, de Vries T, Serruys PW, Samady H, Piek JJ, Lerman A, Escaned J; ADVISE II Study Group. Diagnostic Accuracy of Baseline Distal-to-Aortic Pressure Ratio to Assess Coronary Stenosis Severity: A Post-Hoc Analysis of the ADVISE II Study. JACC Cardiovasc Interv. 2015 May;8(6):834-836. doi: 10.1016/j.jcin.2014.12.245. No abstract available. PMID 25999107
- [Derived] Escaned J, Echavarria-Pinto M, Garcia-Garcia HM, van de Hoef TP, de Vries T, Kaul P, Raveendran G, Altman JD, Kurz HI, Brechtken J, Tulli M, Von Birgelen C, Schneider JE, Khashaba AA, Jeremias A, Baucum J, Moreno R, Meuwissen M, Mishkel G, van Geuns RJ, Levite H, Lopez-Palop R, Mayhew M, Serruys PW, Samady H, Piek JJ, Lerman A; ADVISE II Study Group. Prospective Assessment of the Diagnostic Accuracy of Instantaneous Wave-Free Ratio to Assess Coronary Stenosis Relevance: Results of ADVISE II International, Multicenter Study (ADenosine Vasodilator Independent Stenosis Evaluation II). JACC Cardiovasc Interv. 2015 May;8(6):824-833. doi: 10.1016/j.jcin.2015.01.029. PMID 25999106